CLINICAL TRIAL: NCT03964961
Title: Effect of Functional Massage in Gastrocnemious Muscles Neuromuscular Response
Brief Title: Effect of Functional Massage in Neuromuscular Response.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Principal investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol 6
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-02

CONDITIONS: Neuromuscular Diseases
Keywords: functional massage; conventional massage; neuromuscular response
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The physiotherapist who assesses the outcomes is blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional massage (Experimental)
  Interventions: Other: Functional massage
- Conventional massage (Active Comparator)
  Interventions: Other: Conventional massage

INTERVENTIONS:
Other: Functional massage — It's a massage combined with a stretching of the muscles.
  Arms: Functional massage
Other: Conventional massage — It's a regular massage made with the therapist's hands.
  Arms: Conventional massage

SUMMARY:
The study compares the effects of two types of massage: a conventional massage and a functional massage, in the neuromuscular response of the gastrocnemious muscles.

ELIGIBILITY:
Exclusion Criteria:

* Muscle injury in the last two months
* To not understand the study orders
* Suffer a musculoskeletal disorder that doesn't allow the subject to do the study protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-06-05 (Estimated); Study Completion 2019-06-05 (Estimated)

PRIMARY OUTCOMES:
Delay time change | 2 minutes before the intervention, and 8 minutes after the intervention
  Time between an electric impulse and 10% of the contraction of the muscle that is being excited with an electric impulse, using an electromyography test (miliseconds).
Contraction time change | 2 minutes before the intervention, and 8 minutes after the intervention
  Time between 10% and 90% of the contraction of the muscle that is being excited with an electric impulse, using an electromyography test (miliseconds).
Sustain time change | 2 minutes before the intervention, and 8 minutes after the intervention
  time between 50% of the contraction and 50% of the relaxation of the muscle after being impulsed with an electric impulse, using an electromyography test (miliseconds).
Relaxation time change | 2 minutes before the intervention, and 8 minutes after the intervention
  time between 90% and 50% of the relaxation of the muscle after being impulsed with an electric impulse, using an electromyography test (miliseconds).
Maximal displacement change | 2 minutes before the intervention, and 8 minutes after the intervention
  Maximal displacement of the muscle after being excited with an electric impulse, using an electromyography test (miliseconds).
Stiffness change | 5 minute before the intervention, and 5 minute after the intervention
  Resistance to an external force that deforms its initial shape, using a "Myoton" (N/m).
Elasticity change | 5 minute before the intervention, and 5 minute after the intervention
  Capacity to recover its initial shape after the removal of the external force that lead to its deformation, using a "Myoton" (logarithmic decrement of the tissue's oscillation).
Relaxation change | 5 minute before the intervention, and 5 minute after the intervention
  Time for a muscle to recover its shape from deformation after the removal of an external force, using a "Myoton" (miliseconds).

SECONDARY OUTCOMES:
Gastrocnemious strength change | 8 minutes before the intervention, and 2 minutes after the intervention
  Isometric strength of the gastrocnemious muscles using a handheld dynamometer "microFET 2" (newtons).
Passive ankle dorsiflexion change | 6 minutes before the intervention, and 4 minutes after the intervention
  Passive range of motion of the ankle dorsiflexion, using an inclinometer (degrees).
Jump height change | 10 minutes before the intervention, and 1 minute after the intervention
  Maximum jump height with one leg using the application "My Jump 2" (centimeters).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain